CLINICAL TRIAL: NCT03429894
Title: Evaluation of a Thin Strut Metallic Stent: the Elixir DynamXTM Novolimus Eluting Coronary Bioadaptor System
Brief Title: Evaluation of a Thin Strut Metallic Stent: the Elixir DynamX Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-1704
Record Dates: First submitted 2018-01-17; First posted 2018-02-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: All patients will undergo imaging (angiography and IVUS) follow-up with approximately one-half of the patients returning for follow up at 9 months and approximately one-half returning for follow up at 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All patients will undergo imaging (angiography and IVUS) follow-up with approximately one-half of the patients returning for follow up at 9 months and approximately one-half returning for follow up at 12 months.
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Drug eluting stent implant

SUMMARY:
The DynamX (Bioadaptor) study is a prospective, consecutive enrollment study designed to enroll up to 50 patients requiring treatment of a single, de novo lesion ≤ 24 mm in length located in a vessel ≥ 2.5 mm and ≤ 3.5 mm in diameter. All patients be followed clinically at 30 days, 6 and 9 months, and 1, 2 and 3 years.

All patients will undergo imaging (angiography and IVUS) follow-up with approximately one-half of the patients returning for follow up at 9 months and approximately one-half returning for follow up at 12 months.

DETAILED DESCRIPTION:
The DynamX (Bioadaptor) study is a prospective, consecutive enrollment study designed to enroll up to 50 patients requiring treatment of a single, de novo lesion ≤ 24 mm in length located in a vessel ≥ 2.5 mm and ≤ 3.5 mm in diameter. All patients be followed clinically at 30 days, 6 and 9 months, and 1, 2 and 3 years.

All patients will undergo imaging (angiography and IVUS) follow-up with approximately one-half of the patients returning for follow up at 9 months and approximately one-half returning for follow up at 12 months.

At select centers, a subset of approximately 20 patients will undergo FFR pressure wire measurement at baseline and at follow-up (or at a minimum follow-up) in conjunction with the IVUS imaging, and will also undergo OCT imaging at 9 or 12 months.

The primary safety endpoint is Target Lesion Failure at 6 months. TLF is a composite endpoint defined as cardiac death, target vessel MI, and clinically-indicated target lesion revascularization.

The primary imaging/efficacy endpoints for those patients undergoing imaging follow-up is the change in mean in-device area and mean lumen area at 9 or 12 months compared to post-procedure as measured by IVUS.

Co-primary imaging/efficacy endpoints for those patients undergoing imaging follow-up is late lumen loss as measured by QCA and IVUS at 9 or 12 months.

ELIGIBILITY:
General Inclusion Criteria:

1. Patient must be at least 18 years of age.
2. Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the DynamX Novolimus Eluting Coronary Stent System (CSS) and he/she provides written informed consent, as approved by the appropriate Ethics Committee of the respective clinical site, prior to any clinical study related procedure.
3. Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or electrocardiogram (ECG) changes consistent with ischemia)
4. Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
5. Patient must agree to undergo all clinical study required follow-up visits, angiograms, and IVUS testing
6. Patient must agree not to participate in any other clinical study for a period of one year following the index procedure.

Angiographic Inclusion Criteria - Target Lesion/Vessel

1. Target lesion must be located in a native coronary artery with a nominal vessel diameter of ≥ 2.5 and ≤3.5 mm assessed visually or by online QCA
2. Target lesion must measure ≤ 24 mm in length
3. Target lesion must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 90% with a TIMI flow of ≥ 2
4. The lesion must be successfully pre-dilated (less than 35% DS) prior to enrollment

Angiographic Inclusion Criteria - non-Target Lesion/Vessel Treatment

1. Treatment of a single, non-target lesion located in a separate major epicardial vessel (defined as LAD with septal and diagonal branches, LCX with obtuse marginal and/or ramus intermedius branches and RCA and any of its branches) attempted during the index procedure must be completed first using an approved 'olimus drug eluting stent. The segment must be located such that any injury that might occur during intervention can be clearly attributable to the treated non-target vessel. If the procedure is deemed uncomplicated and optimal, treatment of the target lesion with the DynamX stent can be considered.

Optimal lesion/vessel treatment defined as:

* < 10% but no more than 15% residual diameter stenosis by visual assessment
* no evidence of dissection
* no evidence of thrombus in the treated lesion or vessel
* TIMI 3 flow
* Stent completely covers lesion and extends to healthy vessel on both sides (healthy to healthy)

General Exclusion Criteria

1. Patient has a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure and CK and CK-MB have not returned within normal limits at the time of procedure
2. Patient is currently experiencing clinical symptoms consistent with AMI
3. Patient requires the use of any rotablator intervention during the index procedure
4. Patient has current unstable arrhythmias
5. Patient presenting with heart failure, chronic arrhythmia, COPD or lung function impairment
6. Patient has a known left ventricular ejection fraction (LVEF) < 30%
7. Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
8. Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
9. Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
10. Patient is receiving chronic anticoagulation therapy (e.g., heparin, coumadin) that cannot be stopped and restarted according to local hospital standard procedures.
11. Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel, prasugrel or ticagrelor, Novolimus, CoCr alloys, PLLA polymers or contrast sensitivity that cannot be adequately pre-medicated
12. Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel or other P2Y12 inhibitors.
13. Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease.
14. Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dL, or patient on dialysis)
15. Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
16. Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
17. Patient has had a significant GI or urinary bleed within the past six months
18. Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
19. Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical study plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year)
20. Patient is already participating in another clinical study which has not reached the primary endpoint (long-term follow-up is not an exclusion)
21. Women of childbearing potential who have not undergone surgical sterilization or are not post-menopausal (defined as amenorrheic for at least one year) as well as women who are pregnant or nursing
22. Patient is unable to give their consent, is legally incompetent, or is institutionalized by virtue of an order issued by the courts or other authority

Angiographic Exclusion Criteria

1. Target lesion(s) meets any of the following criteria:

   1. Aorto-ostial location
   2. Left main location
   3. Tapering within target segment of 0.5mm or greater
   4. Located within 10 mm of the origin of the LAD or LCX
   5. Located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
   6. Lesion involving a side branch >2mm in diameter or bifurcation
   7. Previous placement of a stent proximal to or within 10 mm of the target lesion
   8. Total or sub-total occlusion (TIMI flow ≤ 1)
   9. Excessive tortuosity or angulation (≥ 45o) proximal to or within the lesion
   10. The proximal target vessel or target lesion is moderately or severely calcified by visual assessment, or lesion prevents full pre-dilatation balloon expansion
   11. Previous intervention restenosis
2. The target vessel contains visible thrombus
3. Another clinically significant lesion (>40%) is located in the same major epicardial vessel as the target lesion (including side branches)
4. Patient has a high probability that a procedure other than pre-dilatation and stenting and (if necessary) post-dilatation will be required at the time of index procedure for treatment of the target vessel (e.g. atherectomy, cutting balloon)
5. Target vessel was previously treated with any type of PCI < 6 months prior to index procedure
6. Non-Target vessel was previously treated with any type of PCI < 30 days prior to the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 6 months
  Target Lesion Failure (composite of cardiac death, target vessel MI, and clinically-indicated target lesion revascularization)
Change in Mean In-Device Area compared to post-procedure as measured by IVUS | 9 or 12 months
Change in Mean Lumen Area compared to post-procedure as measured by IVUS | 9 or 12 months
Late Lumen Loss (LLL) as measured by QCA | 9 or 12 months
Late Lumen Loss (LLL) as measured by IVUS | 9 or 12 months

SECONDARY OUTCOMES:
Device Success | During Procedure
  Successful delivery of the device and a final residual stenosis < 30% by QCA
Procedure Success | In Hospital through Discharge
  Successful delivery of the device and a final residual stenosis < 30% by QCA without TLF through hospital discharge
Target Lesion Failure (TLF) | 30 days, 1, 2 and 3 years
  Target Lesion Failure (composite of cardiac death, target vessel MI, and clinically-indicated target lesion revascularization)
Cardiac Death | 30 days, 180 days, 1, 2 and 3 years
  Cardiac Death
Non-Cardiac Death | 30 days, 180 days, 1, 2 and 3 years
  Non-Cardiac death
Q-wave Myocardial Infarction (Q-MI) | 30 days, 180 days, 1, 2 and 3 years
  Q-MI
Non-Q-wave Myocardial Infarction (NQ-MI) | 30 days, 180 days, 1, 2 and 3 years
  NQ-MI
Target Vessel Myocardial Infarction (TV-MI) | 30 days, 180 days, 1, 2 and 3 years
  Target Vessel MI
Non-Target Vessel Myocardial Infarction (NTV-MI) | 30 days, 180 days, 1, 2 and 3 years
  Non-Target Vessel MI
Clinically-Indicated Target Lesion Revascularization (CI-TLR) | 30 days, 180 days, 1, 2 and 3 years
  CI-TLR
Non-Clinically Indicated Target Lesion Revascularization (Non-CI-TLR) | 30 days, 180 days, 1, 2 and 3 years
  Non-CI-TLR
Clinically Indicated Target Vessel Revascularization (CI-TVR) | 30 days, 180 days, 1, 2 and 3 years
  CI-TVR
Non-Clinically Indicated Target Vessel Revascularization | 30 days, 180 days, 1, 2 and 3 years
  Non-CI-TVR
Target Vessel Failure (TVF) | 30 days, 180 days, 1, 2 and 3 years
  Composite of cardiac death, target vessel MI, clinically indicated target vessel revascularization
Stent Thrombosis | 30 days, 180 days, 1, 2 and 3 years
  Definite & Probable Stent Thrombosis (per ARC)

OTHER OUTCOMES:
Acute Recoil | During Procedure
  Acute Recoil by QCA
Minimum Lumen Diameter (MLD) | During Procedure
  MLD by QCA
% Diameter Stenosis (DS) | During Procedure
  % DS by QCA
Late Lumen Loss (LLL) | 9 months
  Late lumen loss (in-stent and in-segment) by QCA
Change in mean and minimum lumen, stent and vessel areas from post-procedure | 9 or 12 months
  Change in mean lumen are, device area and vessel area by IVUS
In-stent % neointimal obstruction | 9 or 12 months
  In-stent % neointimal obstruction by IVUS
In-stent late lumen loss (LLL) | 9 or 12 months
  In-stent late lumen loss (LLL) byIVUS
Vasomotion (Pulsatility) | 9 or 12 months
  Vasomotion (Pulsatility) assessment at during systole and diastole by IVUS
Stent malapposition | During procedure, 9 or 12 months
  Acute, persistent and late stent malapposition by IVUS
Fractional Flow Reserve (FFR) | During procedure, 9 or 12 months
  FFR measurements in the treated vessel
Assessment of disengagement segments | 9 or 12 months
  Assessment of disengagement segments by OCT
Incomplete scaffold/device apposition | 9 or 12 months
  Incomplete scaffold/device apposition by OCT
Scaffold/Device Area and Lumen Area | 9 or 12 months
  Scaffold/Device Area and Lumen Area on OCT

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, Principal Investigator — ZNA Middelheim; Antonio Colombo, MD, Principal Investigator — San Raffaele Hospital
Locations (2):
- AZ Middelheim Hospital, Antwerp, Belgium
- Ospendale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Verheye S, Vrolix M, Montorfano M, Giannini F, Bedogni F, Dubois C, De Bruyne B, Costa RA, Chamie D, Costa JR Jr, Abizaid A, Colombo A. Final 36-Month Outcomes from the Multicenter DynamX Study Evaluating a Novel Thin-Strut Novolimus-Eluting Coronary Bioadaptor System and Supporting Preclinical Data. Rev Cardiovasc Med. 2023 Aug 1;24(8):221. doi: 10.31083/j.rcm2408221. eCollection 2023 Aug. PMID 39076703